CLINICAL TRIAL: NCT03902574
Title: A Single Center, Open-label, Randomized, 3-arm, 3-way, Crossover Trial to Investigate the Bioequivalence of Brexpiprazole (OPC-34712) Orally Disintegrating Tablets in Healthy Adult Males
Brief Title: Bioequivalence Study of Brexpiprazole Orally Disintegrating Tablets (ODT) 2mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 331-14-002; JapicCTI-194655 (Other: Japic)
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Healthy Adult Male
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brexpiprazole ODT 2mg with water (Experimental): Brexpiprazole ODT 2mg is administered with water.
  Interventions: Drug: Brexpiprazole ODT 2mg with water
- Brexpiprazole ODT 2mg without water (Experimental): Brexpiprazole ODT 2mg is administered without water.
  Interventions: Drug: Brexpiprazole ODT 2mg without water
- Brexpiprazole conventional tablet 2mg (Experimental): Brexpiprazole conventional tablet 2mg is administered with water.
  Interventions: Drug: Brexpiprazole conventional tablet 2mg

INTERVENTIONS:
Drug: Brexpiprazole ODT 2mg with water — Brexpiprazole ODT 2mg is administered with water.
  Other Names: OPC-34712 OD
  Arms: Brexpiprazole ODT 2mg with water
Drug: Brexpiprazole ODT 2mg without water — Brexpiprazole ODT 2mg is administered without water.
  Other Names: OPC-34712 OD
  Arms: Brexpiprazole ODT 2mg without water
Drug: Brexpiprazole conventional tablet 2mg — Brexpiprazole conventional tablet 2mg is administered with water.
  Other Names: OPC-34712 conventional tablet
  Arms: Brexpiprazole conventional tablet 2mg

SUMMARY:
To investigate the bioequivalence of brexpiprazole ODT 2 mg and brexpiprazole conventional tablet 2 mg

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese males
* BMI ［body weight in kg /(height in m)2］ of at least 18.5 kg/m2 and less than 25.0 kg/m2 (as a result of at the screening examination)
* Capable of providing written informed consent prior to initiation of any trial-related procedures, and able, in the opinion of the investigator, to comply with all requirements of the trial

Exclusion Criteria:

* Clinically significant abnormality at the time of screening (eg, significant deviation from reference ranges) or in medical history that, in the opinion of investigator, subinvestigator, or sponsor may place the subject at risk or interfere with outcome variables such as drug absorption, distribution, metabolism, and excretion
* History of serious mental disorder
* History of drug or alcohol abuse within 2 years prior to screening
* History of any significant drug allergy
* Use of another investigational drug within 120 days prior to the first administration of IMP
* Consumption of grapefruit, grapefruit products, Seville oranges, Seville orange products, Star fruit, or Star fruit products within 72 hours prior to the first administration of IMP or consumption of alcohol within 72 hours prior to administration of IMP
* Use of prescription, over-the-counter (OTC), or herbal medication, or vitamin supplements, or consumption of food or beverages containing St. John's Wort within 14 days prior to the first administration of IMP, or use of antibiotics within 30 days prior to the first administration of IMP
* History of major surgery of the digestive tract (excluding appendectomy)
* Any subject who, in the judgement of the investigator or subinvestigator, should not participate in the trial

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Sato, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- SOUSEIKAI Hakata clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: ODT Without Water/Conventional/ODT With Water: Subjects randomized to Sequence 1 received a brexpiprazole ODT 2 mg without water on Day 1 in Period 1 (Days 1 to 20), then a brexpiprazole conventional tablet 2 mg on Day 21 in Period 2 (Days 21 to 40), then a brexpiprazole ODT 2 mg with water on Day 41 in Period 3 (Days 41 to 60).
- Sequence 2: ODT With Water/ODT Without Water/Conventional: Subjects randomized to Sequence 2 received a brexpiprazole ODT 2 mg with water on Day 1 in Period 1 (Days 1 to 20), then a brexpiprazole ODT 2 mg without water on Day 21 in Period 2 (Days 21 to 40), then a brexpiprazole conventional tablet 2 mg on Day 41 in Period 3 (Days 41 to 60).
- Sequence 3: Conventional/ODT With Water/ODT Without Water: Subjects randomized to Sequence 3 received a brexpiprazole conventional tablet 2 mg on Day 1 in Period 1 (Days 1 to 20), then a brexpiprazole ODT 2 mg with water on Day 21 in Period 2 (Days 21 to 40), then a brexpiprazole ODT 2 mg without water on Day 41 in Period 3 (Days 41 to 60).
Period: Overall Study
Arm/Group | Sequence 1: ODT Without Water/Conventional/ODT With Water | Sequence 2: ODT With Water/ODT Without Water/Conventional | Sequence 3: Conventional/ODT With Water/ODT Without Water
Started | 7 | 7 | 7
Completed | 7 | 7 | 6
Not Completed | 0 | 0 | 1
Not completed — Urinary drug test was positive on Day 20 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set: subjects who received at least one dose of investigational medicinal product (IMP)
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: ODT Without Water/Conventional/ODT With Water | Sequence 2: ODT With Water/ODT Without Water/Conventional | Sequence 3: Conventional/ODT With Water/ODT Without Water | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (6.6) | 27.1 (5.4) | 28.9 (5.4) | 28.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 7 | 7 | 7 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7 | 7 | 7 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 7 | 7 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum (Peak) Plasma Concentration (Cmax) of Brexpiprazole
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12,16, 24, 48, 72, 96, 120, 144, 168, 216, 264 and 312 hours postdose
Population: Bioequivalence analysis set: subjects for whom the relevant bioequivalence variables are available for all periods
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Conventional Tablet: Brexpiprazole conventional tablet 2 mg was administered with water.
- ODT Without Water: Brexpiprazole ODT 2 mg was administered without water.
- ODT With Water: Brexpiprazole ODT 2 mg was administered with water.
Arm/Group | Conventional Tablet | ODT Without Water | ODT With Water
Number analyzed (Participants) | 19 | 19 | 19
ng/mL | 23.31 (4.722) | 24.24 (6.090) | 23.75 (5.320)

2. Primary Outcome: Area Under the Concentration-time Curve Calculated to the Last Observable Concentration at Time t (AUCt) of Brexpiprazole
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12,16, 24, 48, 72, 96, 120, 144, 168, 216, 264, and 312 hours postdose
Population: Bioequivalence analysis set: subjects for whom the relevant bioequivalence variables are available for all periods
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Conventional Tablet | ODT Without Water | ODT With Water
Number analyzed (Participants) | 19 | 19 | 19
ng*h/mL | 1250 (592) | 1340 (629) | 1260 (615)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the start of IMP administration up to 63 days
Description: The safety analysis set consisted of all randomized subjects who received at least one dose of IMP. All the 21 subjects randomized to treatment sequences were included in the safety analysis set.
  (The number of subjects who received conventional tablet, ODT without water, and ODT with water were 21, 20, and 20, respectively).
Arm/Group | Conventional Tablet | ODT Without Water | ODT With Water
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/21 | 2/20 | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Tablet (N=21) | ODT Without Water (N=20) | ODT With Water (N=20)
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Feeling Abnormal (General disorders) | 1 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood Urine Present (Investigations) | 0 | 0 | 1
Dizziness Postural (Nervous system disorders) | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03902574/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03902574/SAP_001.pdf